CLINICAL TRIAL: NCT02148198
Title: A Study of Two Parts to Determine the Effect of NWT-03 on Blood Pressure in Healthy Subjects. Part 1: A Dose Ranging, Cross-over Study to Determine the Effect of 1g, 2g & 5gs of NWT-03 Versus Placebo on Blood Pressure in Healthy Subjects.
Brief Title: Effect of NWT-03 on Blood Pressure - Part 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newtricious R&D BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFCRO-041-part 1
Record Dates: First submitted 2013-11-06; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Blood Pressure
MeSH Terms: interventions — NWT-03

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1g NWT-03, then placebo (Active Comparator): 7 days 1g NWT-03, followed by 7 days placebo, separated by a 5-day wash-out period
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Dietary Supplement: Placebo
- placebo, then 1g NWT-03 (Placebo Comparator): 7 days placebo, followed by 7days 1g NWT-03, separated by a 5-day wash-out period
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Dietary Supplement: Placebo
- 2g NWT-03, then placebo (Active Comparator): 7 days 2g NWT-03, followed by 7 days placebo, separated by a 5-day wash-out period
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Dietary Supplement: Placebo
- placebo, then 2g NWT-03 (Placebo Comparator): 7 days placebo, followed by 7days 2g NWT-03, separated by a 5-day wash-out period
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Dietary Supplement: Placebo
- 5g NWT-03, then placebo (Active Comparator): 7 days 5g NWT-03, followed by 7 days placebo, separated by a 5-day wash-out period
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Dietary Supplement: Placebo
- placebo, then 5g NWT-03 (Placebo Comparator): 7 days 5g NWT-03, followed by 7 days placebo, separated by a 5-day wash-out period
  Interventions: Dietary Supplement: NWT-03, an egg-white protein hydrolysate; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NWT-03, an egg-white protein hydrolysate — For placebo comparator, a combination of sweetener + aroma, which was equal to the combination used in the intervention period, was given
Dietary Supplement: Placebo — A combination of sweetener + aroma, which was equal to the combination used in the intervention period was given as placebo comparator.

SUMMARY:
Part 1 of the study will assess the effect of 1g, 2g and 5g doses of NWT-03 on systolic and diastolic blood pressure in a cross-over designed study in healthy adults with normal, high normal and mild hypertension. Based on results from this study, one dose will be selected for a placebo controlled parallel study assessing a single dose of NWT-03 on systolic and diastolic blood pressure and endothelial function in a similar population.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent,
* Be between 35 and 75 years of age,
* Be in generally good health as determined by the investigator,
* Smokers and non-smokers are eligible,
* Have a stable body weight (< 5% change) over the past 3-months,
* Have a Body Mass Index (BMI) between 25 and 35 kg/m2,
* Be: (a) Normotensive (Systolic Blood Pressure <130 mmHg & Diastolic Blood Pressure <85 mmHg), (b) High normotensive (Systolic Blood Pressure 130-139 mmHg & Diastolic Blood Pressure 85-89 mmHg) or (c) Mild hypertensive (Systolic Blood Pressure 140-159 mmHg & Diastolic Blood Pressure 90-99 mmHg).

Exclusion Criteria:

* Are less than 35 and greater than 75 years of age,
* Females are pregnant, lactating or wish to become pregnant during the study.
* Are hypersensitive to any of the components of the test product,
* Have a significant acute or chronic coexisting illness such as cardiovascular disease, Chronic kidney disease (CKD), gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease or any condition which contraindicates, in the investigators judgement, entry to the study,
* Having a condition or have taken a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include diuretics, blood pressure medication and medication interfering with renin-angiotensin-aldosterone system (RAAS), such as ACE-inhibitors, angiotensin receptor blockers, direct renin inhibitors or aldosterone receptor inhibitor,
* Are taking non-steroidal anti-inflammatory drugs (NSAIDs) within 2 weeks of baseline visit or for the duration of the trial,
* Suffer from diabetes mellitus, either type I and type II,
* Consume more than the recommended alcohol guidelines i.e. >21 alcohol units/week for males and >14 units/week for females,
* History of illicit drug use,
* Use of nasal decongestants and other over-the counter or herbal preparation within 2 weeks of baseline visit and for the duration of the trial,
* Heavy intake of coffee (i.e. more that 4 cups daily) within 2 weeks of baseline visit and for the duration of the trial,
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial,
* Subjects may not be receiving treatment involving experimental drugs,
* If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study. An exception will be made where subjects have participated in part 1 of the study,
* Have a malignant disease or any concomitant end-stage organ disease,

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average daytime systolic blood pressure at 5 days | For both intervention periods: 48h ABPM before baseline visit and 5 days after baseline visit
  Blood pressure will be measured two times for 48h during each intervention period; 48h before the baseline measurement and 5 days after baseline measurement.

SECONDARY OUTCOMES:
Change from baseline in average daytime diastolic blood pressure at 5 days | 48h ABPM before baseline visit and 5 days after baseline visit
  Blood pressure will be measured two times for 48h during each intervention period; 48h before the baseline measurement and 5 days after baseline measurement.
Change from baseline in 48h systolic blood pressure at 5 days | 48h ABPM before baseline visit and 5 days after baseline visit
  Blood pressure will be measured two times for 48h during each intervention period; 48h before the baseline measurement and 5 days after baseline measurement.
Change from baseline in 48h diastolic blood pressure at 5 days | 48h ABPM before baseline visit and 5 days after baseline visit
  Blood pressure will be measured two times for 48h during each intervention period; 48h before the baseline measurement and 5 days after baseline measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Eustace, PhD, Principal Investigator — University College Cork